CLINICAL TRIAL: NCT06063044
Title: Food-specific IgG4-guided Elimination Diets Improve Allergy Symptoms in Children
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: No. 2022-0380
Record Dates: First submitted 2023-06-13; First posted 2023-10-02 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-06

CONDITIONS: Rhinitis, Allergic; Asthma, Allergic; Conjunctivitis, Allergic; Atopic Dermatitis; Chronic Urticaria
Keywords: Immunoglobulin E; Immunoglobulin G; Elimination Diets; chlid
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Conjunctivitis, Allergic; Dermatitis, Atopic; Chronic Urticaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Respiratory system group: the patients who diagnosed as rhinitis, asthma and conjunctivitis were assigned to the respiratory system group
- Skin system group: the patients who diagnosed as urticaria and atopic dermatitis were assigned to the skin system group
- Multiple systems group: the patients who diagnosed with a combination of symptoms from different systems were assigned to the multiple systems group

SUMMARY:
Allergic diseases in children are major public health concerns due to their widespread and rising prevalence. The most classic pathway to trigger allergy is type I allergy mediated by immunoglobulin E(IgE), but the role of immunoglobulin G4(IgG4) in allergic diseases is still worth exploring.we have collected the data of allergic patients aged 0-14 years for retrospective cross-sectional analysis to evaluate the positive rates of total IgE, HDM IgE, FS-IgE and FS-IgG4. Meanwhile, investigators screened out patients who were treated with FS-IgG4-guided elimination diets with/without probiotics for more than 3 months to clarify the role of FS-IgG4 in childhood allergic diseases by assessing the improvement of clinical symptoms before and after treatment.

DETAILED DESCRIPTION:
Allergic diseases in children are major public health concerns due to their widespread and rising prevalence. And management of allergic diseases beyond medication, such as food management is also very important. The most classic pathway to trigger allergy is type I allergy mediated by immunoglobulin E(IgE), but the role of immunoglobulin G4(IgG4) in allergic diseases is still worth exploring.In present study, investigators have collected the data of allergic patients aged 0-14 years for retrospective cross-sectional analysis to evaluate the positive rates of total IgE, house dust mite (HDM) IgE, FS-IgE and FS-IgG4. Meanwhile, investigators screened out patients who were treated with FS-IgG4-guided diet elimination with/without probiotics for more than 3 months to clarify the role of FS-IgG4 in childhood allergic diseases by assessing the improvement of clinical symptoms before and after treatment. This retrospective study was conducted to clarify the clinical relevance of food-specific IgG4 in allergic diseases and the effect of dietary avoidance on clinical symptoms, thus making a breakthrough in the diagnosis and treatment of childhood allergies.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of allergic rhinitis.

* Clinical diagnosis of asthma.
* Clinical diagnosis of conjunctivitis.
* Clinical diagnosis of urticaria.
* Clinical diagnosis of atopic dermatitis.
* Total IgE,FS-IgE, HDM-IgE and FS-IgG4 must be tested.

Exclusion Criteria:

· Autoimmune diseases.

Ages: 8 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A total of 407 patients were recruited. Of the all patients,141 were assigned to the respiratory system group, 124 to the skin system group and 142 to the multiple system group. The follow-up interval of patients in both groups before and after treatment was more than 3 months, with the longest follow-up interval being two and a half years.
Sampling Method: Non-Probability Sample
Enrollment: 407 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Age of participants | 2018.1-2020.12
  Age of participants were evaluated in the respiratory, dermatological and multisystemic groups.
Gender ratio of participants | 2018.1-2020.12
  Gender ratio of participants were evaluated in the respiratory, dermatological and multisystemic groups.
birth mode of participants | 2018.1-2020.12
  Birth mode of participants were evaluated in the respiratory, dermatological and multisystemic groups.
Family history of allergies of the participants | 2018.1-2020.12
  Family history of allergies of the participants were evaluated in the respiratory, dermatological and multisystemic groups.
total IgE | 2018.1-2020.12
  The average level of total IgE in the respiratory, cutaneous, and multi-system groups was assessed.
FS-IgE | 2018.1-2020.12
  The positive rates of FS-IgE in respiratory, cutaneous and multi-system groups were evaluated.
HDM-IgE | 2018.1-2020.12
  The average level of HDM-IgE in the respiratory, cutaneous, and multi-system groups was assessed.
FS-IgG4 | 2018.1-2020.12
  The positive rates of FS-IgG4 in respiratory, cutaneous and multi-system groups were evaluated.
The difference of total-IgE and FS-IgG4 positive rates among the three groups | 2018.1-2020.12
  Chi-square test was used to compare total-IgE (+) FS-IgG4 (+), total-IgE (+) FS-IgG4 (-), total-IgE (-) FS-IgG4 (+) and total-IgE (-) FS-IgG4 (-) among the three groups.
The difference of FS-IgE and FS-IgG4 positive rates among the three groups | 2018.1-2020.12
  Chi-square test was used to compare FS-IgE (+) FS-IgG4 (+), FS-IgE (+) FS-IgG4 (-), FS-IgE (-) FS-IgG4 (+) and FS-IgE (-) FS-IgG4 (-) among the three groups.
Comparison of FS-IgG4 positive rates among the three groups | 2018.1-2020.12
  The differences of 10 food-specific IgG4 antibodies (including eggs, milk, cod, beef, chicken, wheat, prawns, crab, mushrooms) in respiratory, skin and multi-system groups were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Huiying Wang, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Second Affiliated Hospital，School of Medicine，Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No